CLINICAL TRIAL: NCT05950867
Title: Prevalence of Wild-type TTR Cardiac Amyloidosis in Patients With Polyneuropathy of Unknown Cause: a Prospective Monocentric Study (CAP-TTR)
Brief Title: Prevalence of Wild-type TTR Cardiac Amyloidosis in Patients With Polyneuropathy of Unknown Cause.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Veronique Bissay, Principal Investigator, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: EC-2023-115
Record Dates: First submitted 2023-04-21; First posted 2023-07-18 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Polyneuropathy; Amyloidosis
MeSH Terms: conditions — Polyneuropathies; Amyloidosis | interventions — Electrocardiography; Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 1 arm including patients with CAP and/or SFN (Other): 1 arm including patients with chronic axonal length-dependent polyneuropathy and/or small-fiber neuropathy.
  All participants will be screened with ECG and echocardiography. All participants will be asked to complete questionnaires about there polyneuropathy and cardiological symptoms.
  Interventions: Diagnostic Test: ECG + echocardiography; Other: Answering questionnaires

INTERVENTIONS:
Diagnostic Test: ECG + echocardiography — Electrocardiogram and echocardiography
Other: Answering questionnaires — Answering questionnaires about polyneuropathy symptoms (NTSS -6, COMPASS31, NIS, mPND) and also cardialogical symptoms (KCCQ-12).

SUMMARY:
To investigate to what extent chronic axonal length-dependent polyneuropathy (CAP) and/or small-fiber neuropathy (SFN) is part of early non-cardiac manifestations of wild-type TTR cardiac amyloidosis (wtTTR-CA).

Consequently, explore whether this could ultimately lead to faster diagnosis and clinical outcome of wild-type TTR cardiac amyloidosis (wtTTR-CA).

DETAILED DESCRIPTION:
Patients with chronic axonal length-dependent polyneuropathy (CAP) and/or small-fiber neuropathy (SFN) without well-defined cause will be recruited after a neurological standard routine work-up with NCS (Nerve conduction study) test, EMG, and Sudoscan®, previously performed at the neurology department of UZ-Brussel in normal clinical setting. All participants will be invited to the Neurology and Cardiology department for one visit on one day, for the following assessments:

Following exams will be performed:

* assessment of symptoms, severity, and duration of the polyneuropathy and the use of NTSS-6 and COMPASS31 score for mapping somatosensory and autonomic symptoms
* evaluation of objective polyneuropathy signs, using following scales: mPND, NIS
* Kansas City Cardiomyopathy Questionnaire (KCCQ)
* Electrocardiogram (ECG)
* Echocardiography

The following retrospective data from the medical file will be analyzed:

* assessment of medical history, medical treatment, and demographic data
* assessment of laboratory results (and, if applicable, other exams) extracted from the medical file and previously performed in the context of polyneuropathy workup
* assessment of previously performed NCV/EMG data and Sudoscan®, extracted from the medical file of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic axonal length-dependent polyneuropathy (CAP) and/or small-fiber neuropathy (SFN) without well-defined etiology.
* Age: >= 60 years
* Male and female gender
* Written informed consent

Exclusion Criteria:

* Known cause of polyneuropathy
* Other types of peripheral neuropathy than chronic axonal length-dependent polyneuropathy (CAP) and/or small-fiber neuropathy (SFN).
* Patients younger than 60 years

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome: Evaluation of prevalence of wild-type cardiac amyloidosis in our CAP and/or SFN population without well known cause. | 36 months
  Prevalence of cardiac amyloidosis by doing a cardiac screening for wild-type cardiac amyloidosis with performing an echocardiography.
  Echocardiography criteria: LV wall (>12mm), left ventricular ejection fraction (%), Apical sparing pattern (y/n), diastolic dysfunction (y/n), left atrial volume (ml/m2).
  Left atrial volume in ml and LA volume in ml/m2, whereby m2 is the body surface area based on weight and height (Mosteller formula).
Primary Outcome: Evaluation of prevalence of wild-type cardiac amyloidosis in our CAP and/or SFN population without well known cause | 36 months
  Prevalence of cardiac amyloidosis by doing a cardiac screening for wild-type cardiac amyloidosis with performing an ECG.
  ECG criteria: atrial fibrillation (y/n), QRS-duration, low voltage (y/n)
Primary Outcome: Evaluation of prevalence of wild-type cardiac amyloidosis in our CAP and/or SFN population without well known cause | 36 months
  Prevalence of cardiac amyloidosis by doing a cardiac screening for wild-type cardiac amyloidosis with performing a questionnaire (Kansas City Cardiomyopathy Questionnaire).
  KCCQ-12 has 4 domains (Physical Limitation Score, Symptom Frequency Score, Quality of Life Score, Social Limitation Score) and one Summary Score. Scores are scaled 0-100, where 0 denotes the lowest reportable health status and 100 the highest.
  This descriptive score will be used as a functional parameter without a cut-off.

SECONDARY OUTCOMES:
Secondary outcome: severity and evolution | 36 months
  Considering the rather small study population and the rarity of wtTTR amyloidosis, statistical analyses cannot be used without massively overfitting the results, which will not be reproducible. The investigators consequently opt for descriptive statistics to compare the group of polyneuropathy patients with wt-Ca and those without wt-CA. Therefore a few parameters are examined. The first scale used therefore is the modified Polyneuropathy Disability score (mPND). This scale is a questionnaire with a few questions about the complaints of the polyneuropathy in the daily life. O means no complaints of the polyneuropathy in daily life, IV means a major impact on the daily life of the patient.
Secondary outcome: severity and evolution | 36 months
  Considering the rather small study population and the rarity of wtTTR amyloidosis, statistical analyses cannot be used without massively overfitting the results, which will not be reproducible.
  The investigators consequently opt for descriptive statistics to compare the group of polyneuropathy patients with wt-Ca and those without wt-CA. Therefore a few parameters are examined. The second scale used therefore is the Neuropathy Impairment Score (NIS).This scale is a questionnaire with a few questions about the complaints of the polyneuropathy in the daily life. The score is between 0 and 244. O means less complaints in the daily life, 244 means major impact in the daily life of the patient.
Secondary outcome: severity and evolution | 36 months
  Considering the rather small study population and the rarity of wtTTR amyloidosis, statistical analyses cannot be used without massively overfitting the results, which will not be reproducible.
  The investigators consequently opt for descriptive statistics to compare the group of polyneuropathy patients with wt-Ca and those without wt-CA. Therefore a few parameters are examined. The third scale used therefore is the Neuropathy Total Symptom Score - Health Care professional administered version (NTSS-6). This scale is a questionnaire with a few items about the symptoms of the polyneuropathy in the daily life (aching pain, burning pain, prickling sensation, numbness, lancinating pain and allodynia). Depending on the presence of the symptoms in time and strength, a score will show up. On each symptom you can score a maximum of 3,66. So the total score for this scale is 21,96 if the patients has major complaints in daily life.
Secondary outcome: severity and evolution | 36 months
  Considering the rather small study population and the rarity of wtTTR amyloidosis, statistical analyses cannot be used without massively overfitting the results, which will not be reproducible.
  The investigators consequently opt for descriptive statistics to compare the group of polyneuropathy patients with wt-Ca and those without wt-CA. Therefore a few parameters are examined. The fourth scale used therefore is the Composite Autonomic Symptom score (COMPASS-31). This scale is a questionnaire with a 31 questions about the complaints in the daily life and also if there complaints/symptoms on the autonomic system. A few questions are asked about different domains (orthostatic intolerance, vasomotor, secretomotor, gastrointestinal system, bladder, pupillomotor).The total score is minimal 0 and maximal 75 raw counted (100 weighted).Each domain had a weighting factor to be count depending on the answers of the patient.
Secondary outcome: red flags that could increase the awareness of neurologists for wild-type TTR-cardiac amyloidosis | 36 months
  The red flags for wild-type TTR cardiac amyloidosis are among others carpal tunnel syndrome (CTS), wich can be detected by performing an electromyography (EMG).
Secondary outcome: red flags that could increase the awareness of neurologists for wild-type TTR-cardiac amyloidosis | 36 months
  The red flags for wild-type TTR cardiac amyloidosis are among others spinal canal stenosis.
Secondary outcome: red flags that could increase the awareness of neurologists for wild-type TTR-cardiac amyloidosis | 36 months
  The red flags for wild-type TTR cardiac amyloidosis are among others trigger finger.

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Bissay, MD, Phd, Principal Investigator — UZ Brussel - VUB
Locations (1):
- UZ Brussel, Jette, Belgium Capital City, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Russell A, Hahn C, Chhibber S, Korngut L, Fine NM. Utility of Neuropathy Screening for Wild-Type Transthyretin Amyloidosis Patients. Can J Neurol Sci. 2021 Sep;48(5):607-615. doi: 10.1017/cjn.2020.271. Epub 2020 Dec 21. PMID 33342448
- [Background] Kleefeld F, Scherret E, Knebel F, Messroghli D, Heidecker B, Wetz C, Schatka I, Barzen G, Tschope C, Amthauer H, Hahn K. Same same, but different? The neurological presentation of wildtype transthyretin (ATTRwt) amyloidosis. Amyloid. 2022 Jun;29(2):92-101. doi: 10.1080/13506129.2021.2014448. Epub 2022 Jan 7. PMID 34994254
- [Background] Papagianni A, Ihne S, Zeller D, Morbach C, Uceyler N, Sommer C. Clinical and apparative investigation of large and small nerve fiber impairment in mixed cohort of ATTR-amyloidosis: impact on patient management and new insights in wild-type. Amyloid. 2022 Mar;29(1):14-22. doi: 10.1080/13506129.2021.1976751. Epub 2021 Oct 11. PMID 34632904
- [Background] Barroso FA, Coelho T, Dispenzieri A, Conceicao I, Waddington-Cruz M, Wixner J, Maurer MS, Rapezzi C, Plante-Bordeneuve V, Kristen AV, Gonzalez-Duarte A, Chapman D, Stewart M, Amass L; THAOS investigators. Characteristics of patients with autonomic dysfunction in the Transthyretin Amyloidosis Outcomes Survey (THAOS). Amyloid. 2022 Sep;29(3):175-183. doi: 10.1080/13506129.2022.2043270. Epub 2022 Apr 22. PMID 35451899
- [Background] Kharoubi M, Roche F, Bezard M, Hupin D, Silva S, Oghina S, Chalard C, Zaroui A, Galat A, Guendouz S, Canoui-Poitrine F, Hittinger L, Teiger E, Lefaucheur JP, Damy T. Prevalence and prognostic value of autonomic neuropathy assessed by Sudoscan(R) in transthyretin wild-type cardiac amyloidosis. ESC Heart Fail. 2021 Apr;8(2):1656-1665. doi: 10.1002/ehf2.13131. Epub 2020 Dec 22. PMID 33354901
- [Background] Wajnsztajn Yungher F, Kim A, Boehme A, Kleyman I, Weimer LH, Maurer MS, Brannagan TH 3rd. Peripheral neuropathy symptoms in wild type transthyretin amyloidosis. J Peripher Nerv Syst. 2020 Sep;25(3):265-272. doi: 10.1111/jns.12403. Epub 2020 Jul 27. PMID 32627282
- [Background] Zis P, Sarrigiannis PG, Rao DG, Hewamadduma C, Hadjivassiliou M. Chronic idiopathic axonal polyneuropathy: a systematic review. J Neurol. 2016 Oct;263(10):1903-10. doi: 10.1007/s00415-016-8082-7. Epub 2016 Mar 9. PMID 26961897
- [Background] Li Y. Axonal Sensorimotor Polyneuropathies. Continuum (Minneap Minn). 2017 Oct;23(5, Peripheral Nerve and Motor Neuron Disorders):1378-1393. doi: 10.1212/CON.0000000000000514. PMID 28968367
- [Background] Ziemssen T, Siepmann T. The Investigation of the Cardiovascular and Sudomotor Autonomic Nervous System-A Review. Front Neurol. 2019 Feb 12;10:53. doi: 10.3389/fneur.2019.00053. eCollection 2019. PMID 30809183
- [Background] Lehmann HC, Wunderlich G, Fink GR, Sommer C. Diagnosis of peripheral neuropathy. Neurol Res Pract. 2020 Jul 15;2:20. doi: 10.1186/s42466-020-00064-2. eCollection 2020. PMID 33324924
- [Background] England JD, Gronseth GS, Franklin G, Carter GT, Kinsella LJ, Cohen JA, Asbury AK, Szigeti K, Lupski JR, Latov N, Lewis RA, Low PA, Fisher MA, Herrmann DN, Howard JF Jr, Lauria G, Miller RG, Polydefkis M, Sumner AJ; American Academy of Neurology. Practice Parameter: evaluation of distal symmetric polyneuropathy: role of laboratory and genetic testing (an evidence-based review). Report of the American Academy of Neurology, American Association of Neuromuscular and Electrodiagnostic Medicine, and American Academy of Physical Medicine and Rehabilitation. Neurology. 2009 Jan 13;72(2):185-92. doi: 10.1212/01.wnl.0000336370.51010.a1. Epub 2008 Dec 3. PMID 19056666
- [Background] Hanewinckel R, Ikram MA, Van Doorn PA. Peripheral neuropathies. Handb Clin Neurol. 2016;138:263-82. doi: 10.1016/B978-0-12-802973-2.00015-X. PMID 27637963
- [Background] Aimo A, Merlo M, Porcari A, Georgiopoulos G, Pagura L, Vergaro G, Sinagra G, Emdin M, Rapezzi C. Redefining the epidemiology of cardiac amyloidosis. A systematic review and meta-analysis of screening studies. Eur J Heart Fail. 2022 Dec;24(12):2342-2351. doi: 10.1002/ejhf.2532. Epub 2022 May 16. PMID 35509173
- [Background] Gonzalez-Lopez E, Gagliardi C, Dominguez F, Quarta CC, de Haro-Del Moral FJ, Milandri A, Salas C, Cinelli M, Cobo-Marcos M, Lorenzini M, Lara-Pezzi E, Foffi S, Alonso-Pulpon L, Rapezzi C, Garcia-Pavia P. Clinical characteristics of wild-type transthyretin cardiac amyloidosis: disproving myths. Eur Heart J. 2017 Jun 21;38(24):1895-1904. doi: 10.1093/eurheartj/ehx043. PMID 28329248
- [Background] Sperry BW, Reyes BA, Ikram A, Donnelly JP, Phelan D, Jaber WA, Shapiro D, Evans PJ, Maschke S, Kilpatrick SE, Tan CD, Rodriguez ER, Monteiro C, Tang WHW, Kelly JW, Seitz WH Jr, Hanna M. Tenosynovial and Cardiac Amyloidosis in Patients Undergoing Carpal Tunnel Release. J Am Coll Cardiol. 2018 Oct 23;72(17):2040-2050. doi: 10.1016/j.jacc.2018.07.092. PMID 30336828
- [Background] Zegri-Reiriz I, de Haro-Del Moral FJ, Dominguez F, Salas C, de la Cuadra P, Plaza A, Krsnik I, Gonzalez-Lopez E, Garcia-Pavia P. Prevalence of Cardiac Amyloidosis in Patients with Carpal Tunnel Syndrome. J Cardiovasc Transl Res. 2019 Dec;12(6):507-513. doi: 10.1007/s12265-019-09895-0. Epub 2019 Jun 18. PMID 31214980
- [Background] Vianello PF, La Malfa G, Tini G, Mazzola V, Miceli A, Santolini E, Briano S, Porto I, Canepa M. Prevalence of transthyretin amyloid cardiomyopathy in male patients who underwent bilateral carpal tunnel surgery: The ACTUAL study. Int J Cardiol. 2021 Apr 15;329:144-147. doi: 10.1016/j.ijcard.2020.12.044. Epub 2020 Dec 30. PMID 33358831
- [Background] Westin O, Fosbol EL, Maurer MS, Leicht BP, Hasbak P, Mylin AK, Rorvig S, Lindkaer TH, Johannesen HH, Gustafsson F. Screening for Cardiac Amyloidosis 5 to 15 Years After Surgery for Bilateral Carpal Tunnel Syndrome. J Am Coll Cardiol. 2022 Sep 6;80(10):967-977. doi: 10.1016/j.jacc.2022.06.026. PMID 36049804
- [Background] Lindmark K, Pilebro B, Sundstrom T, Lindqvist P. Prevalence of wild type transtyrethin cardiac amyloidosis in a heart failure clinic. ESC Heart Fail. 2021 Feb;8(1):745-749. doi: 10.1002/ehf2.13110. Epub 2020 Nov 17. PMID 33205581
- [Background] Koike H, Okumura T, Murohara T, Katsuno M. Multidisciplinary Approaches for Transthyretin Amyloidosis. Cardiol Ther. 2021 Dec;10(2):289-311. doi: 10.1007/s40119-021-00222-w. Epub 2021 Jun 4. PMID 34089151
- [Background] Maurer MS, Schwartz JH, Gundapaneni B, Elliott PM, Merlini G, Waddington-Cruz M, Kristen AV, Grogan M, Witteles R, Damy T, Drachman BM, Shah SJ, Hanna M, Judge DP, Barsdorf AI, Huber P, Patterson TA, Riley S, Schumacher J, Stewart M, Sultan MB, Rapezzi C; ATTR-ACT Study Investigators. Tafamidis Treatment for Patients with Transthyretin Amyloid Cardiomyopathy. N Engl J Med. 2018 Sep 13;379(11):1007-1016. doi: 10.1056/NEJMoa1805689. Epub 2018 Aug 27. PMID 30145929
- [Background] Campbell CM, LoRusso S, Dispenzieri A, Kristen AV, Maurer MS, Rapezzi C, Lairez O, Drachman B, Garcia-Pavia P, Grogan M, Chapman D, Amass L; THAOS investigators. Sex Differences in Wild-Type Transthyretin Amyloidosis: An Analysis from the Transthyretin Amyloidosis Outcomes Survey (THAOS). Cardiol Ther. 2022 Sep;11(3):393-405. doi: 10.1007/s40119-022-00265-7. Epub 2022 May 18. PMID 35583798
- [Background] Dispenzieri A, Coelho T, Conceicao I, Waddington-Cruz M, Wixner J, Kristen AV, Rapezzi C, Plante-Bordeneuve V, Gonzalez-Moreno J, Maurer MS, Grogan M, Chapman D, Amass L; THAOS investigators. Clinical and genetic profile of patients enrolled in the Transthyretin Amyloidosis Outcomes Survey (THAOS): 14-year update. Orphanet J Rare Dis. 2022 Jun 18;17(1):236. doi: 10.1186/s13023-022-02359-w. PMID 35717381
- [Background] Dyck PJB, Gonzalez-Duarte A, Obici L, Polydefkis M, Wiesman JF, Antonino I, Litchy WJ, Dyck PJ. Development of measures of polyneuropathy impairment in hATTR amyloidosis: From NIS to mNIS + 7. J Neurol Sci. 2019 Oct 15;405:116424. doi: 10.1016/j.jns.2019.116424. Epub 2019 Aug 8. PMID 31445300
- [Background] Bastyr EJ 3rd, Price KL, Bril V; MBBQ Study Group. Development and validity testing of the neuropathy total symptom score-6: questionnaire for the study of sensory symptoms of diabetic peripheral neuropathy. Clin Ther. 2005 Aug;27(8):1278-94. doi: 10.1016/j.clinthera.2005.08.002. PMID 16199253
- [Background] D'Amato C, Greco C, Lombardo G, Frattina V, Campo M, Cefalo CMA, Izzo V, Lauro D, Spallone V. The diagnostic usefulness of the combined COMPASS 31 questionnaire and electrochemical skin conductance for diabetic cardiovascular autonomic neuropathy and diabetic polyneuropathy. J Peripher Nerv Syst. 2020 Mar;25(1):44-53. doi: 10.1111/jns.12366. Epub 2020 Feb 14. PMID 31985124
- [Background] Conceicao I, de Castro I, Castro J. Correlation between Sudoscan and COMPASS 31: assessment of autonomic dysfunction on hATTR V30M patients. Amyloid. 2019;26(sup1):23. doi: 10.1080/13506129.2019.1582494. No abstract available. PMID 31343356